CLINICAL TRIAL: NCT06740409
Title: Accuracy of the Modified Rapid Emergency Medicine Score in Road Traffic Injury: A Prospective Study
Brief Title: Accuracy and External Validation of mREMS in Road Traffic Injuries
Acronym: AVE-MREMS
Status: Recruiting | Type: Observational
Sponsor: Al-Nahrain University (Other)
Responsible Party: Principal Investigator, Abdul-Ilah R. Khamis, Principal Investigator, Al-Nahrain University
Other Study IDs: UNCOMIRB20241214A; 017 (Other: Nahrain Medical Research Collective (NMRC))
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Trauma
Keywords: MREMS
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this prospective observational study is to assess the accuracy and external validation of the Modified Rapid Emergency Medicine Score (mREMS) in predicting outcomes for patients with road traffic injuries (RTIs) admitted to the emergency department of a hospital in Baghdad.

The main questions it aims to answer are:

How accurate is the mREMS in predicting the prognosis of road traffic injury patients? Does the mREMS provide reliable predictive value in a local context, specifically in Baghdad?

Participants will:

Be assessed using the mREMS upon admission to the emergency department. Have their clinical outcomes, including mortality, need for surgery, and length of stay, monitored throughout their hospital stay.

DETAILED DESCRIPTION:
Road traffic injuries (RTIs) are one of the leading causes of morbidity and mortality globally, disproportionately affecting low- and middle-income countries such as Iraq. Accurate and standardized clinical tools are essential for triaging patients and improving clinical outcomes in resource-limited emergency departments. Emergency departments play a central role in the timely assessment and management of RTI patients. The Modified Rapid Emergency Medicine Score (MREMS) has emerged as a valuable tool for predicting in-hospital mortality and other critical outcomes in emergency settings. The Modified Rapid Emergency Medicine Score (mREMS) evaluates key physiological parameters, including age, heart rate, respiratory rate, oxygen saturation, mean arterial pressure, and the Glasgow Coma Scale (GCS), to provide a rapid and standardized assessment of injury severity.

Validation studies in Thailand and other regions have demonstrated mREMS's reliability in predicting in-hospital mortality and critical care needs. These studies have used performance metrics such as sensitivity, specificity, and area under the receiver operating characteristic curve (AUROC) to assess the tool's predictive accuracy. Despite these advancements, there remains a lack of validation studies in Iraq, where healthcare systems face unique challenges, including poor road safety and under-resourced emergency departments.

Previous studies emphasize the importance of adapting and validating scoring systems for specific populations. In Baghdad, RTIs are a significant public health burden, but no standardized tools like mREMS have been validated in this context. This study aims to address this gap by evaluating mREMS's performance in predicting mortality, morbidity, ICU admission, and length of hospital stay requirements in RTI patients in a Baghdad hospital. The findings will contribute to improving trauma care and inform the adaptation of standardized scoring systems in Iraq.

ELIGIBILITY:
Inclusion Criteria:

* Patients with road traffic injuries (RTIs) admitted to the emergency department.
* Written informed consent provided by the patient or a legal representative (if the patient is unconscious or unable to provide consent).
* Patients presenting to the emergency department within 4 hours of the injury.
* Availability of complete physiological data for MREMS calculation.
* Patients whose clinical outcomes (e.g., mortality, length of hospital stay, need for intensive care) are available for follow-up and analysis.

Exclusion Criteria:

* Patients with injuries not related to road traffic accidents (e.g., falls, burns, or violence-related injuries).
* Pregnant women, due to the potential risk involved in the study and unique considerations in trauma care.
* Patients with pre-existing severe chronic conditions (e.g., end-stage renal disease, terminal cancer) that could severely affect outcomes.
* Patients who are unable or unwilling to provide informed consent.
* Patients who were transferred from another hospital.
* Incomplete or missing data for mREMS parameters.
* Patients who leave against medical advice (LAMA) or are discharged before outcome data can be collected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients aged 18 years and older presenting with road traffic injuries (RTIs) to the emergency department of a hospital in Baghdad. These patients will include individuals involved in motor vehicle collisions, motorcycle accidents, pedestrian-related incidents, and other road traffic-related traumas. Participants will be recruited within 4 hours of their injury to ensure timely assessment using the Modified Rapid Emergency Medicine Score (mREMS). Patients with a wide range of injury severities, from minor injuries to life-threatening trauma, will be included to evaluate the score's predictive accuracy across diverse clinical scenarios. The population will be representative of the local demographic and traffic conditions in Baghdad, ensuring the external validation of the mREMS score in this specific context.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
In hospital mortality | In-Hospital Phase (average of 7 days through discharge); Post-Discharge Follow-Up: Day 7, Day 30
  Mortality (death) during hospitalization.
Accuracy Assessment of the modified Rapid Emergency Medicine Score (mREMS) | the first 4 hours after ER admission
  range from 0 to 26. A higher mREMS score indicates a greater risk of mortality.

SECONDARY OUTCOMES:
Length of Hospitalization | Up to discharge, an average of 7 days
  The total duration of a patient's stay in the hospital, measured from the date of admission to the date of discharge. This includes all days spent in general wards, intensive care units (ICU), and other hospital departments as part of their treatment course.
Need for ICU Admission | Up to discharge, an average of 7 days
  The requirement for admission to the intensive care unit (ICU) is determined by the presence of severe clinical deterioration, significant complications, or the need for advanced monitoring and life-support measures.

CONTACTS AND LOCATIONS:
Overall Officials: Bashar A Abdulhassan, Assistant professor of surgery, Study Director — College Of Medicine - Nahrain University
Locations (1):
- College of Medicine - Al-Nahrain University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cassignol A, Markarian T, Cotte J, Marmin J, Nguyen C, Cardinale M, Pauly V, Kerbaul F, Meaudre E, Bobbia X. Evaluation and Comparison of Different Prehospital Triage Scores of Trauma Patients on In-Hospital Mortality. Prehosp Emerg Care. 2019 Jul-Aug;23(4):543-550. doi: 10.1080/10903127.2018.1549627. Epub 2019 Jan 7. PMID 30457396
- [Background] Sewalt CA, Venema E, Wiegers EJA, Lecky FE, Schuit SCE, den Hartog D, Steyerberg EW, Lingsma HF. Trauma models to identify major trauma and mortality in the prehospital setting. Br J Surg. 2020 Mar;107(4):373-380. doi: 10.1002/bjs.11304. Epub 2019 Sep 10. PMID 31503341
- [Result] Miller RT, Nazir N, McDonald T, Cannon CM. The modified rapid emergency medicine score: A novel trauma triage tool to predict in-hospital mortality. Injury. 2017 Sep;48(9):1870-1877. doi: 10.1016/j.injury.2017.04.048. Epub 2017 Apr 25. PMID 28465003
- [Result] Phunghassaporn N, Sukhvibul P, Techapongsatorn S, Tansawet A. Accuracy and external validation of the modified rapid emergency medicine score in road traffic injuries in a Bangkok level I trauma center. Heliyon. 2022 Dec 10;8(12):e12225. doi: 10.1016/j.heliyon.2022.e12225. eCollection 2022 Dec. PMID 36568674